CLINICAL TRIAL: NCT00136240
Title: Telecom System to Improve Adherence to Antidepressants
Brief Title: Automated Telephone System to Improve Treatment Adherence in People With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Ramesh Farzanfar
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: R21MH063937 (NIH); R21MH063937 (NIH); DAHBR HB-A
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2008-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

INTERVENTIONS:
Behavioral: Computer Assisted Education for Behavior Change

SUMMARY:
This study will determine the efficacy of a computerized telephone system called Telephone-Linked Care (TLC) in improving adherence to antidepressant medication regimens in people with depression.

DETAILED DESCRIPTION:
The purpose of this study is to test the efficacy of a computerized telephone system called TLC (Telephone-Linked Care) in helping subjects adhere to their antidepressant medication regimens.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of major depressive disorder, dysthymic disorder, depressive disorder not otherwise specified, or any combination of the three
* Prescribed at least one antidepressant medication
* Access to a telephone with touch-tone service
* Speak and understand conversational English

Exclusion Criteria:

* Current significant alcohol or drug abuse
* Clinical diagnosis of bipolar disorder, schizoaffective disorder, or significant personality disorder
* Parkinson's disease, Huntington's disease, amyotrophic lateral sclerosis (ALS), or other neurodegenerative diseases
* Alzheimer's disease and other dementia
* Cancer, undergoing radiation therapy or chemotherapy
* Suffering from Renal disease or on dialysis
* Immunologic disorder (rheumatoid arthritis, systemic lupus erythematosus [SLE], etc.)
* HIV
* Terminal illness
* Homeless
* Legally blind
* Planning to leave the geographic area during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144
Dates: Start 2003-04; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Antidepressant medication adherence | Measured monthly for 4 months
Adherence to scheduled psychiatry clinic visits | Measured monthly for 4 months

SECONDARY OUTCOMES:
Depression status, measured by self-administered depression inventory scale | Measured at baseline and at 4 month follow-up
General health status, measured by self-rating health survey | Measured at baseline and at 4 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Farzanfar, Study Director — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States